CLINICAL TRIAL: NCT05907746
Title: A Phase II Study of Allogeneic Hematopoietic Stem Cell Transplantation With Briquilimab-Based Conditioning in Participants With GATA2 Deficiency
Brief Title: Allogeneic Hematopoietic Stem Cell Transplantation With Briquilimab-Based Conditioning in Participants With GATA2 Deficiency
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10001531; 001531-C
Record Dates: First submitted 2023-06-15; First posted 2023-06-18 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10-30

CONDITIONS: GATA2; Immunodeficiency
Keywords: Immunodeficiency; Hematopoietic Cell Transplant; Haploidentical
MeSH Terms: conditions — Immunologic Deficiency Syndromes | interventions — Mycophenolic Acid; Tacrolimus; Whole-Body Irradiation; Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Briquilimab, Fludarabine, Total Body Irradiation
  Interventions: Drug: Mycophenolate Mofetil; Drug: Tacrolimus; Drug: Post-Transplant Cyclophosphamide; Radiation: Total Body Irradiation; Procedure: Hematopoietic Cell Transplant; Drug: Briquilimab; Drug: Fludarabine
- Arm B (Experimental): Briquilimab, Fludarabine, Cyclophosphamide, Total Body Irradiation
  Interventions: Drug: Mycophenolate Mofetil; Drug: Tacrolimus; Drug: Post-Transplant Cyclophosphamide; Radiation: Total Body Irradiation; Procedure: Hematopoietic Cell Transplant; Drug: Briquilimab; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Drug: Mycophenolate Mofetil — 15 mg/kg IV three times per day starting on day +5 until approximately day +30 (+/- 2 days)
Drug: Tacrolimus — 0.02 mg/kg IV daily starting on day +5
Drug: Post-Transplant Cyclophosphamide — 50 mg/kg IV daily on days +3 and +4
Radiation: Total Body Irradiation — 200cGy on day -1
Procedure: Hematopoietic Cell Transplant — stem cell transplant on day 0
Drug: Briquilimab — Single 0.6 mg/kg IV infusion administered between days -13 and day -10
Drug: Cyclophosphamide — 14.5 mg/kg IV daily on days -6 and -5; for 7/8 Unrelated or Haploidentical Donor, prior to transplant.
  Arms: Arm B
Drug: Fludarabine — 30 mg/m2 IV over 30 minutes daily. For 8/8 Matched Related or Unrelated Donor, fludarabine dose will be on days -4, -3, and -2. For 7/8 Unrelated or Haploidentical Donor, fludarabine dose will be on days -6, -5, -4, -3, and -2.

SUMMARY:
Background:

People with GATA2 deficiency have a mutation on the GATA2 gene. This gene affects immune function. People with this disease are prone to serious infections; in time, they may develop blood cancers. A hematopoietic stem cell (HSC) transplant can cure GATA2 deficiency, but using stem cells donated by other people can cause serious side effects.

Objective:

To test a new drug (Briquilimab) to see if it can make HSC transplants safer.

Eligibility:

People aged 6 to 70 years who have GATA2 deficiency.

Design:

Participants will be screened. They will have a physical exam, with blood and urine tests. They will have tests of their heart and lung function. They may have a bone marrow biopsy: Their hip will be numbed; a large needle will be inserted to draw out tissue from inside the pelvis.

Participants will have a central venous catheter placed in a vein of the neck or chest. This will be used to draw blood and administer drugs.

Briquilimab will be given through the catheter about 11 days before the transplant. This is part of conditioning: preparing the body to receive the new stem cells. Conditioning also includes other medications and total body irradiation.

Donor stem cells will be administered through the catheter. Participants will receive other approved drugs to help prevent side effects.

Participants will stay in the hospital from the beginning of the conditioning until several weeks after the transplant. They will remain in the local area for 100 days after discharge; they will come to the clinic at least once a week during this time. Follow-up visits will continue for 3 years....

DETAILED DESCRIPTION:
Background:

* GATA2 deficiency, an immunodeficiency and bone marrow failure disorder due to inherited or sporadic mutations in or loss of one allele of the GATA2 gene, is characterized by: 1) nontuberculous mycobacteria (NTM) and other opportunistic infections, 2) deficiency of monocytes, B lymphocytes, and Natural Killer (NK) cells in the peripheral blood, and 3) progression to myelodysplastic syndrome (MDS), chronic myelomonocytic leukemia (CMML), and acute myelogenous leukemia (AML).
* Allogeneic hematopoietic cell transplantation (HCT) appears to be curative, and interim results from protocol #13-C-0132, NCT01861106, demonstrated a 2-year event-free survival rate of 83% for 59 participants with GATA2 deficiency who underwent HCT with a busulfan-based conditioning regimen.
* However, traditional HCT approaches using alkylating agents such as busulfan continue to place recipients at risk for potentially life-threatening, transplant-related toxicities as well as late effects such as infertility and secondary malignancy.
* Briquilimab is a humanized, glycosylated IgG1 monoclonal antibody that targets CD117 (human c-Kit) present on endogenous hematopoietic stem cells (HSC). Briquilimab has been shown in pre-clinical and early clinical studies to safely deplete human and non-human primate HSC with minimal toxicity.

Primary Objective:

-To determine whether allogeneic hematopoietic cell transplantation with Briquilimab-based conditioning results in sustained donor engraftment by 100 days post-transplant in participants with GATA2 deficiency

Eligibility:

* Recipients aged 6-70 years old with pathogenic germline mutations in GATA2 and clinical manifestations consistent with a diagnosis of GATA2 deficiency
* Have an 8/8 Human leukocyte antigen (HLA)-matched related or unrelated donor or a 7/8 HLA-matched unrelated donor or haploidentical related donor
* Have "early stage" GATA2 deficiency defined as a hypocellular for age bone marrow with less than 5% blasts and normal or favorable cytogenetics (defined as "good" or "very good" cytogenetics risk groups plus trisomy 8)

Design:

* All participants with GATA2 deficiency will receive a pre-transplant conditioning regimen consisting of Briquilimab administered as a single intravenous (IV) infusion on day -11 (range day -13 to -10) with pharmacokinetics, followed by fludarabine or fludarabine/cyclophosphamide IV infusions (3 or 5 days depending on the donor) and 200 cGy total body irradiation (TBI) on day -1. HCT will be infused on day 0.
* Participants with an 8/8 HLA-matched related or unrelated donor assigned to Arm A will receive a fludarabine for three days on days -4, -3, and -2.
* Participants with a 7/8 HLA-matched unrelated donor or a haploidentical related donor assigned to Arm B will receive a fludarabine for five days on days -6, -5, -4, -3, and -2, cyclophosphamide for 2 days on days -6 and -5
* Post-transplant immunosuppression for Graft Versus Host Disease (GVHD) prophylaxis for recipients of Arms A and B will consist of cyclophosphamide for 2 days on days +3 and +4, along with mycophenolate mofetil from day +5 to approximately day +35 and tacrolimus from day +5 to approximately day +180. If there is no evidence of GVHD, tacrolimus will be stopped or tapered at approximately day +180

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age >= 6 and <= 70 years old
* Germline mutation in the GATA2 gene, predicted to be deleterious or previously reported in GATA2 deficiency as determined by targeted GATA2 sequencing performed at the NIH
* Clinical manifestation(s) consistent with a diagnosis of GATA2 deficiency, including any of the following (Note: only one clinical manifestation is required):

  * History of severe, disfiguring, and/or recurrent infections
  * Low monocyte (< 190 cells/microL), B cell (< 61 cells/microL) and/or NK cell (< 126 cells/microL) counts
  * Myelodysplastic syndrome by World Health Organization (WHO) criteria
* "Early stage" GATA2 deficiency defined as a hypocellular for age bone marrow with less than 5% blasts and normal cytogenetics or favorable cytogenetics (defined as "good" or "very good" cytogenetics risk groups plus trisomy 8)
* Availability of an 8/8 HLA-matched related or unrelated donor, a 7/8 HLA-matched unrelated donor or a haploidentical related donor
* Lansky (for participants < 16 years of age) or Karnofsky (for participants >=16 years of age) performance status of >= 40%
* Left ventricular ejection fraction > 40%, preferably by 2-D echocardiogram (echo) obtained within 90 days prior to treatment initiation
* Participants must have adequate organ function as defined below:

  * Total bilirubin <=2.5 x upper limit of normal (ULN)
  * Alanine transaminase (ALT) and aspartate aminotransferase (AST) <= 5 x ULN
  * Creatinine:

Adult participants: <=2.0 mg/dl and creatinine clearance >= 30 ml/min.

Pediatric participants (<18 years old): creatinine <1.5 mg/dL and a creatinine clearance using the Schwartz Formula > 30 mL/min/1.73m^2

* Pulmonary function tests (PFT)s: FEV1 and adjusted DLCO >30%. Children who are unable to cooperate for PFTs due to age are still eligible if no evidence of dyspnea at rest and no need for supplemental oxygen
* Women of childbearing potential (WOCBP) and men must agree to use highly effective contraception (hormonal, intrauterine device (IUD), abstinence, tubal ligation, partner has had the previous vasectomy) at the study entry, for the duration of study treatment, and for at least one-year post-allogeneic HCT or 12 months after completion of chemotherapy preparative administration if HCT is not performed for women and for 4 months for the same for men.
* Breastfeeding participants must be willing to discontinue breastfeeding
* Willingness to remain in the NIH hospital or, if discharged, stay close to the NIH (60 minutes drive), for a minimum of 100 days after transplant or longer if there are complications. The participants must commit to having an adult caregiver with them during the first 100 days after transplant in case of discharging from the hospital before 100 days verified by social worker
* Participants with hepatitis B virus (HBV) or hepatitis C virus (HCV) antibody-positive testing are allowed if HBV DNA <100 IU/m or HCV RNA level is undetectable. Additionally, transplantation must be approved by a hepatology consult for these participants
* Participants or parents/guardians must be able to understand and willing to sign a written informed consent document

EXCLUSION CRITERIA:

* Participants with a Hematopoietic Cell Transplantation-Comorbidity Index (HCT-CI) score >8
* Participants who have received any investigational agents within 4 weeks before treatment initiation with the exception of virus-specific T cells for the treatment of viral infection/reactivation prior to allogeneic HCT
* Participants with a history of hematologic malignancy (e.g., AML, CMML). Note: participants with MDS are included
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to agents (fludarabine, cyclophosphamide, tacrolimus, mycophenolate mofetil, granulocyte-colony stimulating factor (G-CSF)) used in the study
* Presence of active malignancy. Note: participants with malignancy driven by viruses (e.g., human papillomavirus (HPV) or HPV or Epstein-Barr virus (EBV)) are allowed as the immune reconstitution after transplant may control the malignancy and participants with MDS are allowed
* Human immunodeficiency virus (HIV)-infected participants
* Pregnancy (confirmed with Beta-HCG serum or urine pregnancy test performed in WOCBP at screening)
* Uncontrolled intercurrent illness or social situations (as determined by social work consult) that would limit compliance with study requirements

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-11-29 (Actual); Primary Completion 2025-10-16 (Actual); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
To determine whether allogeneic hematopoietic cell transplantation with Briquilimab-based conditioning results in sustained donor engraftment by 100 days post-transplant in participants with GATA2 deficiency | 100 days post-transplant
  Fraction of evaluable participants reported along with one-sided 90% confidence intervals and a two-sided 95% confidence interval

SECONDARY OUTCOMES:
To determine whether allogeneic hematopoietic cell transplantation with Briquilimab-based conditioning results in restoration of normal hematopoiesis by one-year post-transplant in participants with GATA2 deficiency | 1 year post-transplant
  Fraction of evaluated participants reported along with a 95% two-sided confidence interval.
The safety of allogeneic HCT in participants with GATA2 deficiency conditioned with Briquilimab | 3 years post-transplant
  By arm, the participants with transplant-related toxicity will be reported by type and grade of event.
3-year overall survival | 3 years post-transplant
  Determined using the Kaplan-Meier method, along with the median value and the 95% confidence interval
3-year event-free survival | 3 years post-transplant
  Determined using the Kaplan-Meier method, along with the median value and the 95% confidence interval
3-year incidence of secondary graft failure | 3 years post-transplant
  Fraction of participants will be reported separately by cohort along with 95% two-sided confidence interval
3-year incidence of grade III-IV acute and moderate to severe chronic graft versus host disease | +1, +2, and +3 years post-transplant
  Fractions of participants will be reported separately by cohort using simple estimates along with 95% two-sided confidence intervals. In addition, cumulative incidence curves along with 95% two-sided confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle E Pregent-Arnold, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001531-C.html